CLINICAL TRIAL: NCT00392288
Title: A Multicenter, Multi-national, Randomized, Double-blind, Placebo-controlled, Study to Assess the Efficacy and Safety of Ciclesonide Metered-dose Inhaler (MDI) at 80 μg BID or 40 μg BID for 12 Weeks in Patients Aged 4 to <12 Years With Persistent Asthma.
Brief Title: Efficacy and Safety of Ciclesonide (CIC) Administered Twice Daily in Pediatric Patients With Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6695; XRP1526
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo MDI (Placebo Comparator): double-blind
  Interventions: Drug: Placebo
- Ciclesonide MDI 40 µg BID (Experimental): double-blind
  Interventions: Drug: Ciclesonide
- Ciclesonide MDI 80 µg BID (Experimental): double-blind
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: Ciclesonide — Ciclesonide MDI 40 µg BID over twelve weeks
  Arms: Ciclesonide MDI 40 µg BID
Drug: Ciclesonide — Ciclesonide MDI 80 µg BID over twelve weeks
  Arms: Ciclesonide MDI 80 µg BID
Drug: Placebo — Placebo MDI over twelve weeks
  Arms: Placebo MDI

SUMMARY:
Primary objective: To demonstrate the efficacy of ciclesonide, compared to placebo, at 80 μg twice daily (BID) or 40 μg BID for 12 weeks in patients with persistent asthma.

Secondary objective: To assess the safety and tolerability of ciclesonide.

ELIGIBILITY:
Inclusion Criteria:

* History of persistent bronchial asthma for at least 3 months prior to screening;
* For patients with persistent bronchial asthma and being treated with a controller therapy: Documented use of an inhaled steroid or Singulair® 5mg once daily;
* For patients with persistent bronchial asthma and not being treated with controller therapy: Patients may have documented use of a reliever therapy such as albuterol/salbutamol or may be untreated;
* Morning Peak Expiratory Flow (AM PEF) of ≤90% of predicted values from the in-clinic spirometry after a 6 hour withhold of albuterol/salbutamol;
* Only patients aged between 6 to <12 years must have a forced expiratory volume in one second (FEV1) of ≥50% to ≤85% of predicted normal after a 6 hour withhold of albuterol/salbutamol

Exclusion Criteria:

* Nocturnal awakenings for asthma which require treatment with albuterol/salbutamol for 4 or more nights out of the last 7 days of the screening period;
* Use of more than 8 puffs/day of albuterol/salbutamol on 3 or more consecutive days within the last 7
* Upper or lower respiratory tract infection within 4 weeks prior to screening and during screening period;
* History of life-threatening asthma, including a history of significant hypercarbia (pCO2 >45 mmHg), prior intubation, respiratory arrest, or seizures as a result of an exacerbation of asthma;
* More than 3 in-patient hospitalization or emergency care visits due to asthma exacerbations in the year prior to screening;
* Use of injectable or oral corticosteroids within one month prior to screening, or more than 3 bursts) within 6 months prior to screening;

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (6):
- sanofi-aventis, US, Bridgewater, New Jersey, United States
- Sanofi-Aventis Hungaria, Budapest, Hungary
- Sanofi-Aventis, México, Mexico
- sanofi-aventis Poland, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Moscow, Russia
- sanofi-aventis South Africa, Midrand, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening period 7-14 days, randomization with subsequent treatment period over 12 weeks
Pre-assignment Details: The number of subjects in section Participant Flow is related to the number of randomized subjects (= subject who were eligible for treatment period). This number is different to the number of subjects of the Intention to Treat (ITT) population in Outcome Measures. The statistical analyses of the Outcome Measures is related to the ITT population.
Groups:
- Placebo Metered Dose Inhaler (MDI): Placebo MDI over twelve weeks (ITT population)
- Ciclesonide MDI 40 µg BID: Ciclesonide MDI 40 µg BID over twelve weeks (ITT population)
- Ciclesonide MDI 80 µg BID: Ciclesonide MDI 80 µg BID over twelve weeks (ITT population)
Period: Overall Study
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID
Started | 175 (Number of randomized subjects is different to number of ITT population in Outcome Measures.) | 177 (Number of randomized subjects is different to number of ITT population in Outcome Measures.) | 176 (Number of randomized subjects is different to number of ITT population in Outcome Measures.)
Treatment Period | 172 | 174 | 175
Completed | 143 (ITT set = 163 patients) | 155 (ITT set = 166 patients) | 159 (ITT set = 172 patients)
Not Completed | 32 | 22 | 17
Not completed — Adverse Event | 17 | 7 | 8
Not completed — Lack of Efficacy | 8 | 5 | 3
Not completed — Protocol Violation | 1 | 3 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Parent/legal guardian withdrawal | 1 | 2 | 1
Not completed — Other | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID | Total
Number analyzed (Participants) | 163 | 166 | 172 | 501
Age, Customized [Number; unit: participants]
  Aged 6 to <12 years | 136 | 138 | 145 | 419
  Aged 4 to <6 years | 27 | 28 | 27 | 82
Gender [Count of Participants; unit: Participants]
  Female | 59 | 70 | 75 | 204
  Male | 104 | 96 | 97 | 297

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Week 12.
Description: Change in FEV1 (Percent of predicted) from baseline to week 12. FEV1 was measured only in children between 6 to <12 years only. Least Squares Mean were adjusted for Baseline FEV1, age [yrs], pooled center, previous corticosteroid therapy and holding chamber.
Time Frame: Baseline and Week 12
Population: Analyses are based on children of the ITT population. It includes all randomized patients who have a baseline and a valid post-randomization lung function measurement. The primary analysis was restricted to an age range between 6 and <12 years.
Measure: Least Squares Mean (Standard Error); unit: Percent of predicted FEV1
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID
Number analyzed (Participants) | 136 | 138 | 146
Percent of predicted FEV1 | 5.2 (1.06) | 5.3 (1.06) | 7.7 (1.06)
Statistical Analysis 1: Comparison: Placebo Metered Dose Inhaler (MDI) vs Ciclesonide MDI 40 µg BID vs Ciclesonide MDI 80 µg BID; This is an analysis of the change from baseline to week 12 or last visit. In this pairwise comparison Ciclesonide was compared with Placebo by testing the average effect of Ciclesonide 40 and Ciclesonide 80 versus Placebo. As statistical test a t-test was used to compare the corresponding least-square means of both treatment groups; Test type: Superiority or Other; p = 0.2696, ANCOVA — Due to usage of a-priori ordered hypotheses, adjustment of p-values is not necessary. The pre-specified significance level was 0.05. The tests were carried out two-sided; ANCOVA model: Change in FEV1 = baseline FEV1 + age [yrs] + treatment + pooled center + previous corticosteroid therapy + holding chamber
Statistical Analysis 2: Comparison: Placebo Metered Dose Inhaler (MDI) vs Ciclesonide MDI 80 µg BID; This is an analysis of the change from baseline to week 12 or last visit. A t-test was used to compare the least-square means of Ciclesonide 80 versus Placebo; Test type: Superiority or Other; p = 0.0703, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo Metered Dose Inhaler (MDI) vs Ciclesonide MDI 40 µg BID; This is an analysis of the change from baseline to week 12 or last visit. As statistical test a t-test was used to compare the corresponding least-square means of Ciclesonide 40 versus Placebo; Test type: Superiority or Other; p = 0.9146, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Total Daily Asthma Symptom Score at Week 12.
Description: Change in total daily asthma symptom score from baseline to week 12. 5-Point, ordinal scale specifying patient's experience of symptoms during day and night from 0 (no symptoms) to 4 (symptoms that prevent the patient from engaging in daily activities or sleep)
Time Frame: Baseline and Week 12
Population: Analyses are based on children of the ITT population. It includes all randomized patients who have a baseline and a valid post-randomization lung function measurement.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID
Number analyzed (Participants) | 161 | 165 | 170
Scores on a scale | -0.96 (0.08) | -1.13 (0.08) | -0.99 (0.08)

3. Secondary Outcome: Change From Baseline in Use of Albuterol/Salbutamol at Week 12.
Description: Change in albuterol/salbutamol use from baseline to week 12
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Puffs per day
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID
Number analyzed (Participants) | 162 | 166 | 172
Puffs per day | -0.59 (0.08) | -0.87 (0.08) | -0.93 (0.08)

ADVERSE EVENTS:
Description: The numbers of subjects at risk are based on the Safety Population. It was based on all randomized patients receiving at least one dose of the double-blind study medication after randomization.
Arm/Group | Placebo Metered Dose Inhaler (MDI) | Ciclesonide MDI 40 µg BID | Ciclesonide MDI 80 µg BID
Serious Adverse Events (participants affected / at risk) | 1/172 | 1/174 | 4/175
Other Adverse Events (participants affected / at risk) | 53/172 | 38/174 | 28/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Metered Dose Inhaler (MDI) (N=172) | Ciclesonide MDI 40 µg BID (N=174) | Ciclesonide MDI 80 µg BID (N=175)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Forearm fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Electric shock (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Metered Dose Inhaler (MDI) (N=172) | Ciclesonide MDI 40 µg BID (N=174) | Ciclesonide MDI 80 µg BID (N=175)
Headache (Nervous system disorders) | 5 (5) | 12 (18) | 8 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 10 (10) | 3 (3)
Nasopharyngitis (Infections and infestations) | 9 (11) | 8 (9) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 4 (5) | 10 (10)
Pharyngitis (Infections and infestations) | 17 (19) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days